CLINICAL TRIAL: NCT02013635
Title: Study of Thrombin Generation and Thrombus Degradation in Cerebral Venous Thrombosis : Correlation With Clinical and Radiological Evolution
Brief Title: Thrombin Generation and Thrombus Degradation in Cerebral Venous Thrombosis : Clinical and Radiological Correlations
Acronym: PHRC-TVC
Status: Completed | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2010/087/HP
Record Dates: First submitted 2011-11-28; First posted 2013-12-17 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-11

CONDITIONS: Cerebral Venous Thrombosis
Keywords: cerebral venous thrombosis; thrombin generation; d-dimers; clinical evolution
MeSH Terms: conditions — Intracranial Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — plasma, serum and whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cerebral Venous Thrombosis: patients over 16 years old with acute cerebral venous thrombosis

SUMMARY:
Cerebral venous thrombosis is considered as a rare type of stroke with an annual incidence of 3 to 4 per million people. It occurs generally in young patients (mean age of occurrence = 40 years) and principally in young females (75%) generally in pregnancy or oral contraceptive use situations.

The onset may be acute (less than 2 days), subacute (between 2 and 30 days) or chronic (more than 30 days). The clinical presentation is highly variable and includes patients with only a mild headache, others with focal neurological deficits and a few with a dramatic syndrome and a coma. Moreover the evolution can be very different with unpredictable outcome: more often it is favorable with a low mortality rate, but in some cases it can be a worse course. The aim of this study is to evaluate the correlation of some biological markers: thrombin generation test and D-Dimers (marker of fibrin generation and degradation) with the type of onset or the wide spectrum of clinical presentations or the different modes of evolution.

All patients over 16 years ago may be included in the program when CVT diagnosis is proved by magnetic resonance angiography (MRA). For each included patient, there are four blood assays: the first just at the time of diagnosis and before the beginning of treatment, the second before the beginning of the oral anticoagulant treatment. The third assay is done in the third month at the time of a MRA. The last assay is made one month after the end of the anticoagulant treatment or in 12th month after the beginning of the disease if the treatment goes on.

For each sample, the investigators perform a thrombin generation test and a D-Dimers measurement.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 16 years old hospitalized with an acute cerebral venous thrombosis, confirmed by by cerebral imaging

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients over 16 years old hospitalized with an acute cerebral venous thrombosis
Sampling Method: Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2011-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evolution of thrombin generation parameters | one year
  Evolution from Baseline in thrombin generation parameters and correlation with clinical presentation (initial state and severity with NIH stroke scale and GLASGOW Scale)
Evolution of D Dimers concentration | one year
  Evolution from Baseline in D Dimers concentration and correlation with clinical presentation (initial state and severity with NIH stroke scale and GLASGOW Scale)

SECONDARY OUTCOMES:
Evolution of thrombin generation parameters after end of treatment | one year
  Evolution from end of treatment in thrombin generation parameters and correlation with clinical presentation (initial state and severity with NIH stroke scale and GLASGOW Scale)
MR Imaging and Thrombin generation parameters | one year
  Number of venous occlusions on MR Imaging and correlation with thrombin generation parameters
MR Imaging and D Dimers concentration | one year
  Number of venous occlusions on MR Imaging and correlation with D Dimers concentration
Evolution of D Dimers concentration after treatment | one year
  Evolution from end of treatment in D Dimers concentration and correlation with clinical presentation (initial state and severity with NIH stroke scale and GLASGOW Scale)

CONTACTS AND LOCATIONS:
Overall Officials: LE CAM DUCHEZ VERONIQUE, MD, Study Director — CHU HOPITAUX DE ROUEN
Locations (36):
- France (36):
  - Chu Amiens, Amiens
  - Chu D' Angers, Angers
  - Ch Victor Dupouy, Argenteuil
  - CH Côte Basque, Bayonne
  - Hôpital Jean Minjioz, Besançon
  - Hôpital Pellegrin - CHU Bordeaux, Bordeaux
  - Hôpital de la Cavale Blanche, Brest
  - Hôpital Neurologique de Lyon, Bron
  - Hôpital Côte de Nacre, Caen
  - CHU Estaing, Clermont-Ferrand
  - Hôpitaux Civils de Colmar, Colmar
  - C.H. de Compiègne, Compiègne
  - Hôpital Henri Mondor, Créteil
  - CHU-Hôpital Général, Dijon
  - C.H.I. Eure-Seine, Évreux
  - C.H.U. de Grenoble, Grenoble
  - C.H. de La Rochelle, La Rochelle
  - C.H. de Versailles, Le Chesnay
  - Hôpital J. Monod, Le Havre
  - C.H.U. Limoges, Limoges
  - C.H. François Quesnay, Mantes-la-Jolie
  - Hôpital de la Timone, Marseille
  - C.H. de Meaux, Meaux
  - Hôpital Guy de Chauliac, Montpellier
  - Hôpital Nord de Laënnec, Nantes
  - G.H.U. Carémeau, Nîmes
  - G.H. Paris Saint-Joseph, Paris
  - GH Pitié-Salpêtrière, Paris
  - C.H. de Perpignan - Hôpital Saint-Jean, Perpignan
  - CHI de Poissy- site de Poissy, Poissy
  - C.H.U de Poitiers, Poitiers
  - CHU hopitaux de rouen, Rouen
  - C.H. Yves Le Foll, Saint-Brieuc
  - C.H. Saint-Denis, Saint-Denis
  - C.H.U de Strasbourg, Strasbourg
  - CHRU Bretonneau, Tours

REFERENCES:
- [Derived] Triquenot Bagan A, Crassard I, Drouet L, Barbieux-Guillot M, Marlu R, Robinet-Borgomino E, Morange PE, Wolff V, Grunebaum L, Klapczynski F, Andre-Kerneis E, Pico F, Martin-Bastenaire B, Ellie E, Menard F, Rouanet F, Freyburger G, Godeneche G, Allano HA, Moulin T, Mourey G, Derex L, Berruyer M, Runavot G, Trichet C, Viader F, Le Querrec A, Husein TT, Cluet-Dennetiere S, Macian-Montoro F, Donnard M, Guillon B, Ternisien C, Zuber M, Laplanche S, Tassan P, Peeltier JY, Canaple S, Roussel B, Gaillard N, Scavazza E, Le Cam Duchez V. Cerebral Venous Thrombosis: Clinical, Radiological, Biological, and Etiological Characteristics of a French Prospective Cohort (FPCCVT)-Comparison With ISCVT Cohort. Front Neurol. 2021 Nov 8;12:753110. doi: 10.3389/fneur.2021.753110. eCollection 2021. PMID 34819911